CLINICAL TRIAL: NCT04487171
Title: Screening for Postpartum Depression and Associated Risk Factors Among Women Who Deliver in Four Hospital in France During the COVID-19 Epidemic
Acronym: COVIE-19/20
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Beauvais (Other); Central Hospital Saint Quentin (Other Government); Centre Hospitalier Compiègne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0049
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Postpartum Depression; Covid19; Prevalence; Social Distance
Keywords: Postpartum Depression; Covid19; Prevalence; Social Distance
MeSH Terms: conditions — Depression, Postpartum; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The mothers were administrated three questionnaires, (i) the Edinburgh Postnatal Depression Scale (EPDS), (ii) the State-Trait Anxiety Inventory (STAI-YA), and (iii) the Mother-to-Infant Bonding Scale (MIBS) in two stages, on days 2-3 after delivery and during a phone call between days 25-35.

SUMMARY:
Postpartum depression (PPD) represent around 15% of birth in developed countries. The context of the COVID-19 epidemy represents a possible source of additional emotional distress. The objective of this study is to determine the screening prevalence and risk factors of postpartum depression, among women who deliver in fourth hospital in the North of France in the context of the COVID epidemy.

ELIGIBILITY:
Inclusion Criteria:

* Single baby delivery
* alive new born child without admission in neonatal intensive care unit
* French-speaking mother
* mother older than 18 years old

Exclusion Criteria:

* Patients who refuses the inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women who deliver
Enrollment: 248 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Variation of prevalence of clinically-significant post-partum depressive symptoms | up to 35 days after delivery
  Variation of prevalence of clinically-significant post-partum depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Arthur FOULON, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No